CLINICAL TRIAL: NCT04788433
Title: ROCCO - Registry of Coronavirus Complications. Prospective Observational Study on Coronavirus Complications and Correlation With Glycomic Profile in COVID-19 Patients
Brief Title: Registry of Coronavirus Complications - CORRELATION WITH GLYCOMIC PROFILE in COVID-19 Patients
Acronym: ROCCO
Status: Completed | Type: Observational
Sponsor: Papa Giovanni XXIII Hospital (Other)
Collaborators: GENOS (Other)
Responsible Party: Principal Investigator, Dario Bugada, Anesthesiologist, Papa Giovanni XXIII Hospital
Other Study IDs: ROCCO-197/2020
Record Dates: First submitted 2021-03-07; First posted 2021-03-09 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain; Morbidity, Multiple; Covid19
MeSH Terms: conditions — Chronic Pain; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- ROCCO-A (A-symptomatic): Patients with documented COVID-19 infection and NO symptoms
  Interventions: Diagnostic Test: glycomic analysis; Other: Phone interview
- ROCCO-P (Pauci-symptomatic): Patients with documented COVID-19 infection and mild symptoms but NO oxygen support)
  Interventions: Diagnostic Test: glycomic analysis; Other: Phone interview
- ROCCO-L (mild): Patients with documented COVID-19 infection and mild severity - requiring OXIGEN SUPPORT
  Interventions: Diagnostic Test: glycomic analysis; Other: Phone interview
- ROCCO-M (moderate): Patients with documented COVID-19 infection and moderate severity - requiring OXIGEN SUPPORT by NON-INVASIVE modalities
  Interventions: Diagnostic Test: glycomic analysis; Other: Phone interview
- ROCCO-S(severe): Patients with documented COVID-19 infection and severe disease requiring INVASIVE VENTILATION OR EXTRACORPOREAL MEMBRANE OXYGENATION
  Interventions: Diagnostic Test: glycomic analysis; Other: Phone interview

INTERVENTIONS:
Diagnostic Test: glycomic analysis — Analysis of glycans on plasma samples
Other: Phone interview — patients are followed up by phone up to 1 year

SUMMARY:
COVID infection has resulted in multi-organ injury and may result in cardiovascular, pulmonary, neurological, and muscular damage. It is associated with significant asthenia and the long-term effects of the infection are still unclear, particularly for the development of pain and delayed functional rehabilitation.

Glycomics "is the systematic study of the structure of glycans in a given cell type or organism. Glycans are complex oligosaccharides attached to proteins and lipids that regulate a variety of organic processes, including immunity Thus, glycans may influence different moments of the response to the virus and involved in the clinical severity of the disease, but may also change depending on the severity of symptoms and the organic response to SARS-CoV-2 infection.

Glycomic data could provide important insights into interindividual differences at the molecular level that directly interact with SARS-CoV-2 and the development of mid- and long-term side effects. The ability to identify early those susceptible to developing COVID-19 infection and at higher risk for COVID-19 with unfavorable outcomes long after infection would help guide therapeutic strategy and provide important guidance for rational health care organization, which is of outmost importance.

Long-term outcome data regarding post-COVID patient functional capacity and glycomics will be compared to assess whether there may be differences in protein glycosylation that may predict patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID19 virus infection (buffer/BAL/positive IgG serology)
* Age >18 years
* Able to express informed consent to participate in the study

Exclusion Criteria:

* patients unable to express consent,
* patients aged <18 yr,
* with signs and symptoms compatible with Covid-19 but without certified diagnosis by swab/BAL or serological examination of presence of COVID IgG antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented infection by Sars-CoV2 with different degrees of clinical severity.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Glycomic profile as predictor of long-term morbidity | 1 year
  Analysis of total plasmatic and IgG glycans composition; analysis of IgG glycopeptides. Correlation with pain, severity of the disease and long-term functional rehabilitation

CONTACTS AND LOCATIONS:
Locations (1):
- Aast Papa Giovanni Xxiii, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No